CLINICAL TRIAL: NCT04209166
Title: A Study of Individualized Diagnosis and Treatment for Major Depressive Disorder With Atypical Features
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: Air Force Military Medical University, China (Other); Guangzhou Psychiatric Hospital (Other Government); Dalian Seventh People's Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CRC2018ZD05
Record Dates: First submitted 2019-12-16; First posted 2019-12-23 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-10

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Selective Serotonin Reuptake Inhibitors; Serotonin and Noradrenaline Reuptake Inhibitors; Serotonin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- FAD (Experimental): the first-episode major depressive disorder with atypical feature
  Interventions: Drug: SSRIs/SNRIs (Selective Serotonin Reuptake Inhibitors/ Serotonin and Norepinephrine Reuptake Inhibitors); Drug: SSRIs/SNRIs+Mood Stabilizer; Drug: SSRIs/SNRIs+Quetiapine; Drug: Usual Treatment
- RAD (Experimental): the recurrent major depressive disorder with atypical feature who have been medication-free for no less than 2 weeks
  Interventions: Drug: SSRIs/SNRIs (Selective Serotonin Reuptake Inhibitors/ Serotonin and Norepinephrine Reuptake Inhibitors); Drug: SSRIs/SNRIs+Mood Stabilizer; Drug: SSRIs/SNRIs+Quetiapine; Drug: Usual Treatment
- BD (No Intervention): the depressive episode of bipolar disorder
- HC (No Intervention): healthy control

INTERVENTIONS:
Drug: SSRIs/SNRIs (Selective Serotonin Reuptake Inhibitors/ Serotonin and Norepinephrine Reuptake Inhibitors) — Patients will be treated with Selective Serotonin Reuptake Inhibitors/ Serotonin and Norepinephrine Reuptake Inhibitors.
  Arms: FAD; RAD
Drug: SSRIs/SNRIs+Mood Stabilizer — Patients will be treated with Mood Stabilizer combined with Selective Serotonin Reuptake Inhibitors/ Serotonin and Norepinephrine Reuptake Inhibitors.
  Arms: FAD; RAD
Drug: SSRIs/SNRIs+Quetiapine — Patients will be treated with Quetiapine combined with Selective Serotonin Reuptake Inhibitors/ Serotonin and Norepinephrine Reuptake Inhibitors.
  Arms: FAD; RAD
Drug: Usual Treatment — Patients' treatment will be decided by the clinical doctor.
  Arms: FAD; RAD

SUMMARY:
The lifetime prevalence of major depressive disorder (MDD) is 10%~20%. Worldwide, nearly 340 million individuals have suffered the torture of depression. World Health Organization has reported that MDD would become the most serious global burden of disease and eventually turn into a public health problem in 2030. Varied clinical symptoms, inappropriate treatment, unclear pathogenesis, and lack of recurrent risk early-warning predictors cause a series of clinical problems, such as low diagnostic rate, low effective treatment rate, and high recurrent rate. Hence, this study aims to search multidimensional markers for early diagnosis of MDD, to establish optimized personalized therapy, and to explore sensitive recurrence predictors.

Based on the criteria of the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5), MDD is subdivided into eight different clinical specifiers, one of which the incident rate of MDD with atypical features reaches 30%~38%. However, there is still a lack of meta-evidence for the clinical treatment strategy in MDD with atypical features. And 45.4 percentage of MDD with atypical features convert to bipolar disorder. Therefore, this study will focus on three issues about what's the objective endophenotype in MDD with atypical features, how to select appropriate personalized treatment for MDD with atypical features, what's the predictive biomarker of conversion to bipolar disorder.

Based on the investigators' previous findings, this study will investigate adult depression at a cross-sectional study and a prospective cohort study. Multivariate informatics analysis was performed from three research dimensions (cognitive neuropsychology, metabonomics, and multimodal neuroimaging), including atypical features, "cold/hot" cognition assessment, KP (kynurenine pathway) metabolomics and inflammatory factors, multimodal MRI robust property. Referring guidelines for the diagnosis and treatment of depression and evidence-based medicine evidence, MDD with atypical features are divided into f groups (antidepressants, antidepressants+mood stabilizers, mood stabilizers, treat as usual). Then, the investigators perform follow-up to verify optimized treatment strategies and to explore risk factors of conversion from MDD with atypical features to bipolar disorder. Furthermore, this study performs correlation analysis to analyze cross-omics data, weight coefficient analysis to analyze multidimensional indexes, clustering analysis to analyze multivariate bio-information data, and artificial intelligence technologies (such as pattern recognition, and machine learning) to realize the transformation from medical data to practical transformation. Eventually, this study builds three specific models (the multidimensional early diagnosis models for MDD with atypical features, the optimized personalized therapy model, and the recurrence and conversion risk early-warning model), which form the integrated intelligent platform for multidimensional diagnosis, personalized treatment, recovery management of MDD with atypical features.

ELIGIBILITY:
Inclusion Criteria:

1. 16-60 years old;
2. Meeting with the criteria of major depressive disorder in the Diagnostic and Statistical Manual of Mental Disorders (DSM)-5;
3. Scored 20 or higher on the Hamilton's Depression Scale with 24 items (HAMD-24);
4. With enough audio-visual ability and comprehensive ability to accomplish the visits;
5. Be necessary and suitable to accept the treatment of antidepressants;
6. Scored less than 14 on Hamilton's Anxiety Scale (HAMA) and scored less than 14 on the Hypomania Symptom Checklist-32 (HCL-32);
7. With 2 or more atypical symptoms including significant weight gain or increase in appetite, hypersomnia, leaden paralysis, and a long-standing pattern of interpersonal rejection sensitivity that results in significant social or occupational impairment.

Exclusion Criteria:

1. Severe medical or neurological problems;
2. Previous mania or hypomania episodes;
3. Female patients who are pregnant, planning to be pregnant or breastfeeding;
4. Actively suicide ascertained by research psychiatrist or 3rd item of HAMD scored≥3(suicidality);
5. Had ECT, MECT or rTMS in the past 6 months;
6. Experienced severe personality disorder, mental retardation, anorexia/bulimia nervosa.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 780 (Estimated)
Dates: Start 2019-08-12 (Actual); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
remission of acute phase | 12th week
  scored 7 or lower on the Hamilton's Depression Scale with 24 items
switch rate | 4th year
  the rate of patients who switch from depression to mania or hypomania during 4-year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Daihui Peng, MD. PhD., Study Chair — Shanghai Mental Health Center
Locations (5):
- China (5):
  - Guangzhou Psychiatric Hospital, Guanzhou, Guangdong
  - Wuhan Mental Health Center, Wuhan, Hubei
  - Dalian Seventh People's Hospital, Dalian, Liaoning
  - Shanghai Mental Health Center, Shanghai, Shanghai Municipality
  - Fourth Military Medical University, Xian, Shanxi

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhou R, Zhang H, He S, Li Y, Xu G, Huang J, Wang H, Wang Q, Li B, Wang X, Chen N, Li F, Li X, Liu M, Peng D. A Study of Individualized Diagnosis and Treatment for Depression with Atypical Features (iDoT-AFD): study protocol for a randomized clinical trial and prognosis study. Trials. 2023 May 4;24(1):308. doi: 10.1186/s13063-023-07317-w. PMID 37143128